CLINICAL TRIAL: NCT07404280
Title: Intervention of Artificial Intelligence in the Management of Nutritional Therapy Applied to Moroccan Type 2 Diabetics - Al-Khawarizmi Project
Brief Title: Impact of a Nutritional Intervention Based on Moroccan Dietary Habits on the Glycemic Control of Type 2 Diabetics
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Avicenna Military Hospital (Other)
Responsible Party: Principal Investigator, Zineb Kabbaj, PhD student, Avicenna Military Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 153/2024/2026
Record Dates: First submitted 2026-02-05; First posted 2026-02-11 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Type 2 Diabetes (T2DM)
Keywords: Type 2 Diabetes; Artificial Intelligence; Nutritional Intervention; Glycemic Control; Moroccan Dietary Habits; Precision Nutrition
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Adapted Nutritional Intervention (Experimental): A single group of 50 Type 2 Diabetic patients will participate in a four-stage intervention over 180 days.
  * Phase 1 (Baseline): Participants will follow their usual, free diet for 7 days while monitored by Continuous Glucose Monitoring (CGM) and food diaries to establish a baseline.
  * Phase 2 (Intervention): Participants receive personalized nutritional directives specifically adapted to traditional Moroccan dietary habits and culinary practices.
  * Phase 3 (Follow-up): Continuous monitoring and periodic consultations (at Day 14, Day 90, and Day 180) to adjust the intervention, measure metabolic changes (HbA1c), and evaluate anthropometric parameters.
  Interventions: Behavioral: Moroccan-Adapted Nutritional Plan

INTERVENTIONS:
Behavioral: Moroccan-Adapted Nutritional Plan — The intervention consists of a structured diet plan that integrates traditional Moroccan ingredients and cooking methods while optimizing for glycemic control. It involves:
  * Personalized meal planning based on individual food diaries.
  * Education on carbohydrate counting and portion sizes within the Moroccan culinary context.
  * Use of Continuous Glucose Monitoring (CGM) data to provide real-time feedback on how specific Moroccan meals affect the participant's glucose levels.

SUMMARY:
The goal of this study is to learn if a nutritional intervention adapted to Moroccan dietary habits can improve blood sugar control in adults with Type 2 Diabetes. The main questions it aims to answer are:

* Does a personalized diet based on Moroccan culinary traditions improve long-term blood sugar levels (HbA1c)?
* How does this intervention affect daily blood sugar fluctuations measured as interstitial glucose?
* Does the intervention lead to changes in body measurements, such as weight and Body Mass Index (BMI)?

Participants will:

* Wear a Continuous Glucose Monitor (CGM) to track sugar levels in real-time.
* Keep a detailed food diary of all foods and drinks consumed.
* Follow their usual diet for the first 7 days to establish a baseline.
* Receive personalized dietary advice specifically tailored to Moroccan food habits.
* Return for clinical check-ups at 14, 90, and 180 days for blood tests and body measurements.

DETAILED DESCRIPTION:
This study follows a quasi-experimental, before-after design conducted in a clinical setting. The research is structured to evaluate the metabolic and anthropometric response of Type 2 Diabetic (T2D) patients to a culturally tailored nutritional intervention. The trial is longitudinal, spanning a total duration of 180 days per participant.

Intervention Phases:

The protocol is divided into distinct chronological stages to capture both baseline data and intervention outcomes:

* Baseline Phase (Days 1-7): Participants maintain their habitual "free" diet to establish a baseline for glycemic variability and caloric intake. During this phase, Continuous Glucose Monitoring (CGM) systems and detailed food diaries are used to map postprandial glucose responses to traditional Moroccan meals.
* Intervention Initiation (Day 7- T7): A specialized dietitian analyzes the baseline food diaries and CGM cycles to provide personalized nutritional directives. These directives adapt international dietary standards to the specific ingredients, cooking methods, and flavor profiles of Moroccan cuisine.
* Adjustment and Stabilization (Day 14- T14): A follow-up consultation is held to assess initial adherence and refine the nutritional recommendations based on the participant's feedback and early glycemic data.
* Medium and Long-term Follow-up (T90 & T180): Metabolic stability is evaluated at 3 and 6 months. These stages involve comprehensive biological testing and anthropometric measurements to determine the sustainability of the intervention's effects.

Data collection and Scientific tools:

The study utilizes high-precision monitoring tools to ensure data reliability:

* Continuous Glucose Monitoring (CGM): Sensors are used to record interstitial glucose levels in real-time, providing a more granular view of glycemic control that traditional finger-stick testing.
* Nutritional Analysis: Food intake is quantified through structured diaries, kitchen scales for portion control, and validated food frequency questionnaires.
* Anthropometric and metabolic Markers: Bioelectrical impedance analysis (BIA) is used to track body composition changes, while laboratory tests measure HbA1c, fasting blood glucose, and lipid and renal profiles.

Statistical Analysis Plan Data will be analyzed using a within-subject comparison. Descriptive statistics will summarize baseline characteristics. Paired t-tests and ANOVA will be employed to compare glycemic and anthropometric variables across the four time points (T0, T7, T90, T180), with a significance level set to p<0.05. Additionally, Pearson or Spearman correlation tests and Artificial Intelligence techniques will examine the association between specific Moroccan dietary patterns and glycemic fluctuations.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of T2D by a healthcare professional.
* Age 18 years or older.
* A glycated hemoglobin (HbA1c) level less than 10%.
* Capacity to provide informed written consent and follow the study procedures.

Exclusion Criteria:

* Non-diabetic subjects.
* Type 1 diabetes or secondary diabetes.
* Age younger than 18 years.
* Pregnancy or planned pregnancy during the study period.
* HbA1c level greater than 10%.
* Chronic renal insufficiency or hepatic disease.
* Pathologies of the digestive tract that affect nutrient absorption.
* Known food allergies requiring highly specific restricted diets.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Change in Interstitial Glucose Levels | Baseline (Day 0 to Day 7) compared to the final follow-up at Day 180.
  Evaluation of the impact of the Moroccan-adapted nutritional intervention on daily glucose fluctuations. This is measured using a Continuous Glucose Monitoring (CGM) system to record real-time glucose data.

SECONDARY OUTCOMES:
Change in HbA1c | Baseline (Day 0) and Day 180.
  Measurement of glycated hemoglobin to assess long-term glycemic control through laboratory samples.
Change in Body Mass Index (BMI) | Baseline (Day 0) and Day 180.
  Calculation of BMI based on weight and height measurements.
Change in Waist Circumference | Baseline (Day 0) and Day 180.
  Anthropometric measurement of the waist to evaluate changes in abdominal adiposity.
Change in Body Composition | Baseline (Day 0) and Day 180.
  Assessment of body fat and lean mass using bioelectrical impedance.
Dietary Adherence | Baseline (Day 7) compared to Day 180.
  Evaluation of changes in dietary habits and adherence to the personalized Moroccan-adapted recommendations using food diaries.

CONTACTS AND LOCATIONS:
Overall Officials: Hicham Baïzri, Study Director — Department of Endocrinology, Diabetology and Metabolic Diseases, Avicenne Military Hospital, Marrakech, Morocco
Locations (1):
- Avicenna Military Hospital of Marrakech, Marrakesh, Marrakech Safi, Morocco

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this study and the final article (text, tables, figures, and appendices), after de-identification, will be made available to researchers who provide a methodologically sound proposal. Request should be directed to the corresponding author. To gain access, data requestors will need to sign a data access agreement.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available beginning 6 months after publication of the results and ending 3 years after publication.
Access Criteria: Data will be shared with researchers who provide a methodologically sound proposal and after signing a data access agreement to ensure ethical use and patient anonymity.